CLINICAL TRIAL: NCT02683252
Title: Magnetic Resonance (MR) Imaging Quantitative Functional Perfusion Analysis of the Musculoskeletal System: Clinical Application in Non-tumoral Pathology
Brief Title: Musculoskeletal Non-tumoral Pathology Quantitative Perfusion
Acronym: AFRONT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RCB: 2015-A01604-45
Record Dates: First submitted 2016-01-28; First posted 2016-02-17 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Osteonecrosis; Pseudarthrosis; Compartment Syndrome
Keywords: Magnetic resonance imaging; perfusion; quantitative
MeSH Terms: conditions — Osteonecrosis; Pseudarthrosis; Compartment Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Normal patients (Experimental): Patients with normal bone appearance on conventional MR images
  Interventions: Other: T1 mapping and MR perfusion acquisition
- Carpal osteonecrosis (Experimental): Patients presenting signal anomalies compatible with osteonecrosis of the carpal bones on conventional MR images (hypointensity on T1 weighted sequences, no contrast enhancement).
  Interventions: Other: T1 mapping and MR perfusion acquisition
- Femoral head osteonecrosis (Experimental): Patients presenting signal anomalies compatible with osteonecrosis of the femoral head on conventional MR images (fat containing signal anomalies with geographic contours in the femoral epiphysis).
  Interventions: Other: T1 mapping and MR perfusion acquisition
- Pseudarthrosis (Experimental): Patients presenting a non consolidated macroscopic bone fracture for over 6 months (clinical history and imaging findings).
  Interventions: Other: T1 mapping and MR perfusion acquisition
- Compartment syndrome (Experimental): Patients with a confirmed compartment syndrome on intra-compartment pressure assessement
  Interventions: Other: T1 mapping and MR perfusion acquisition

INTERVENTIONS:
Other: T1 mapping and MR perfusion acquisition — One T1 mapping acquisition with variable flip angles will be performed before contrast injection. One perfusion 3D FSPGR sequence will be acquired after contrast injection

SUMMARY:
Study on quantitative perfusion parameters acquired on MR imaging of patients with non-tumoral pathology of the musculoskeletal system.

DETAILED DESCRIPTION:
Patients referred for the MR imaging evaluation of non-tumoral musculoskeletal pathology (osteonecrosis, pseudarthrosis and compartment syndrome) will have their MR protocols complemented by a contrast enhanced perfusion study. In this patients standard clinical evaluation is already performed with contrast medium injection (Gadolinium) and no additional injection is required.

After post processing multiple quantitative perfusions parameters will be extracted (e.g. plasmatic volume, transfer constant, backflow constant, extra-cellular extra vascular space volume). The variation of these parameters in patients with and without the previously described conditions will be compared.

ELIGIBILITY:
Inclusion Criteria:

* affiliation to a social security regimen
* Signature of an informed consent
* Clinical suspicion of one of the studied conditions (osteonecrosis of the wrist, osteonecrosis of the femoral head, pseudarthrosis and compartment syndrome)

Exclusion Criteria:

* MR contraindications
* Contraindications to contrast injection
* Previous history of allergy to gadolinium containing contrast medium
* Presence of metallic hardware in the study zone
* Pregnancy
* Patients under tutelage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-02-12 (Actual); Primary Completion 2019-02-12 (Estimated); Study Completion 2020-02-12 (Estimated)

PRIMARY OUTCOMES:
Variation of the plasmatic volume estimation in the 5 study groups (arms) and between the images acquired in the two inclusion sites. | 3 years
  The plasmatic volume (Vp%) in ml is a quantitative perfusion parameter that describes the capillar density of the tissues evaluated and can be useful in tissue characterization

SECONDARY OUTCOMES:
Variation of the plasma-extra-cellular space transfer constant in the 5 study groups (arms) and between the images acquired in the two inclusion sites. | 3 years
  The plasma-extracellular space transfer constant (Ktrans) in min -1 is a quantitative perfusion parameter that is related to the capillar permeability and blood flow. This parameter can be useful for tissue characterization.
Variation of the extra-cellular space-plasma transfer constant (backflow constant) in the 5 study groups (arms) and between the images acquired in the two inclusion sites. | 3 years
  The extracellular-space-plasma transfer constant or backflow constant (Kep) in min -1 is a quantitative perfusion parameter that is related to the capillar permeability. This parameter can be useful for tissue characterization.
Variation of the extra-cellular extra-vascular space volume in the 5 study groups (arms) and between the images acquired in the two inclusion sites. | First 6 months of inclusion
  The extracellular-space extra-vascular space volume (Ve%) in ml is a quantitative perfusion parameter that is related to the tissue cellularity. This parameter can be useful for tissue characterization.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CCIAL, CHRU-Lille, Lille, Hauts-de-France
  - Service d'Imagerie Guilloz, CHRU-Nancy, Nancy, Lorraine

REFERENCES:
- [Background] Mueller D, Schaeffeler C, Baum T, Walter F, Rechl H, Rummeny EJ, Woertler K. Magnetic resonance perfusion and diffusion imaging characteristics of transient bone marrow edema, avascular necrosis and subchondral insufficiency fractures of the proximal femur. Eur J Radiol. 2014 Oct;83(10):1862-9. doi: 10.1016/j.ejrad.2014.07.017. Epub 2014 Jul 30. PMID 25129825
- [Background] Muller GM, Mansson S, Muller MF, Ekberg O, Bjorkman A. Assessment of perfusion in normal carpal bones with dynamic gadolinium-enhanced MRI at 3 Tesla. J Magn Reson Imaging. 2013 Jul;38(1):168-72. doi: 10.1002/jmri.23951. Epub 2012 Nov 27. PMID 23188589
- [Background] Bervian MR, Ribak S, Livani B. Scaphoid fracture nonunion: correlation of radiographic imaging, proximal fragment histologic viability evaluation, and estimation of viability at surgery: diagnosis of scaphoid pseudarthrosis. Int Orthop. 2015 Jan;39(1):67-72. doi: 10.1007/s00264-014-2579-4. Epub 2014 Nov 16. PMID 25398469
- [Background] Rominger MB, Lukosch CJ, Bachmann GF. MR imaging of compartment syndrome of the lower leg: a case control study. Eur Radiol. 2004 Aug;14(8):1432-9. doi: 10.1007/s00330-004-2305-5. Epub 2004 Apr 6. PMID 15067424
- [Result] Teixeira PA, Chanson A, Beaumont M, Lecocq S, Louis M, Marie B, Sirveaux F, Blum A. Dynamic MR imaging of osteoid osteomas: correlation of semiquantitative and quantitative perfusion parameters with patient symptoms and treatment outcome. Eur Radiol. 2013 Sep;23(9):2602-11. doi: 10.1007/s00330-013-2867-1. Epub 2013 May 22. PMID 23695220